CLINICAL TRIAL: NCT05627713
Title: Description of the Kinetics of the Clinical and Biological Aspects of the Persons Consulting in the Framework of the Management of the MONKEYPOX Disease
Brief Title: Clinical and Biological Aspects of the MONKEYPOX Disease
Acronym: PoxVac22
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Centre Médical de l'Institut Pasteur (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-078; 2022-A01915-38 (Other: ID-RCB)
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Monkey Pox
Keywords: vaccination; infection; monkey pox virus; outbreak; immunization
MeSH Terms: conditions — Mpox, Monkeypox; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals coming to CMIP for MONKEYPOX disease management (Other): * 300 individuals eligible for MPXV vaccination and
  * 30 individuals suspected of MPXV infection.
  Interventions: Other: Blood sample collection; Other: urine sample collection

INTERVENTIONS:
Other: Blood sample collection — Blood sample collection between inclusion and 12 months after inclusion
Other: urine sample collection — urine sample collection at inclusion

SUMMARY:
Monkey pox virus (MPXV), of the genus Orthopoxvirus, regularly causes epidemics in endemic areas of central and western Africa.

Since January 1, 2022, cases of Monkey pox have been reported to WHO by 96 Member States in the 6 WHO regions. As of 22 August 2022, a total of 41,664 laboratory-confirmed cases and 192 probable cases, including 12 deaths, have been reported to WHO. Since May 13, 2022, a high proportion of these cases have been reported from countries where monkey pox transmission had not previously been documented. For the first time, cases and sustained chains of transmission are being reported in countries without direct or immediate epidemiological links to areas in West or Central Africa (WHO 2022). France is one of the most affected countries with 2889 cases reported as of August 22, 2022.

This situation led the WHO Director General to declare, on July 23, 2022, that the monkeypox epidemic currently affecting several countries constitutes a Public Health Emergency of International Concern.

To address this epidemic, the WHO has recommended Post Exposure Vaccination (PEP) and Pre Exposure Vaccination (PrEP) for at risk groups with 2nd and 3rd generation vaccines. In France, the Haute Autorité de Santé (French National Authority for Health) recommended on May 20, 2022, vaccination for PEP and on July 7, 2022, for PrEP with a 3rd generation MVA-BN vaccine (Imvanex® or Jynneos®). The European Medicines Agency (EMA) has approved the use of Imvanex® on July 22, 2022 for immunization against MPXV.

The objective of the present study is to describe the clinical, biological, virological, pathophysiological and immunological aspects in the short and medium term of persons vaccinated against and infected with MPXV.

DETAILED DESCRIPTION:
Descriptive, prospective, monocentric, longitudinal study. Subjects will be enrolled during their consultation at CMIP as part of their curative or preventive management of MPXV disease.

At the time of the appointment dedicated to vaccination or as part of the diagnosis of the infection, the clinician will explain the study in progress and will propose to the individual to participate if he/she is eligible.

If so, after signing the informed consent form, the individual will be included in the study.

The collection of socio-demographic, clinical and treatment data will be done on an eCRF at each study visit.

Biological samples (blood and/or urine samples and/or swabs for viruses) will also be taken at each study visit.

The samples will be used for the following biological analyses

* serological analyses
* sero-neutralization analysis by different techniques
* cytometric analyses and biomarker measurements
* virological analyses
* genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult,
* eligible for MPXV vaccination according to HAS criteria or suspected of MPXV infection
* whose health status is compatible with a 45 ml single blood sample
* who have consented to participate in the study
* who are covered by a Social Health Insurance plan

Exclusion Criteria:

* Person with MPXV vaccination without proof of vaccination.
* For persons presenting for MPXV vaccination: presence of a contraindication to vaccination other than a current infection.
* Pregnant and lactating women
* Person unable to give informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Characterize the immune responses of the individual to MPXV vaccination | 5 years
  Seroneutralizing capacity of serum 14 days (+/- 2 days) after the last dose administered
Characterize the developed cellular immunity and circulating levels of immune signaling molecules in individuals after MPXV vaccination and MPXV infection | 5 years
  Measurement of activation of dendritic cells, NK cells, B cells and various T cells and levels of involved cytokines in individuals after MPXV vaccination and MPXV infection
Map the presence of MPXV in infectious sites of infected patients by qualitative and quantitative analyses comparing primary lesions, secondary lesions and healthy skin | 5 years
  Measurement of the number of clinical sites in which MPXV is demonstrated, the level of associated viral load, the cellular distribution of lesional viral load on biopsies of ulcerated areas
Characterize gene expression profiling in the peripheral blood of the individual after MPXV vaccination and the individual after MPXV infection | 5 years
  Transcriptomic analysis of gene expression of immunological markers in individuals after MPXV vaccination and MPXV

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Taieb, MD, Principal Investigator — Institut Pasteur
Locations (1):
- Centre Médical de l'Institut Pasteur, Paris, France